CLINICAL TRIAL: NCT04043962
Title: Mechanisms Of Change in Adolescent Pain Self-management
Acronym: MOCAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Tonya Palermo, Professor, Anesthesiology and Pain Medicine, Seattle Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R21NR017312 (NIH)
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Results first posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-09

CONDITIONS: Chronic Pain; Central Sensitisation; Headache
Keywords: chronic pain; internet intervention; pain management; CBT; adolescent; sleep
MeSH Terms: conditions — Chronic Pain; Headache; Agnosia

STUDY DESIGN:
Intervention Model Description: All participants will receive internet-delivered CBT for pain self-management (Web-MAP).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Web-based CBT (Web-MAP) (Experimental): The eight child modules include: 1) education about chronic pain, 2) recognizing stress and negative emotions, 3) deep breathing and relaxation, 4) implementing coping skills at school, 5) cognitive skills (e.g., reducing negative thoughts), 6) lifestyle interventions, 7) staying active (e.g., pleasant activity scheduling), 8) relapse prevention. The eight parent modules are: 1) education about chronic pain, 2) recognizing stress and negative emotions, 3) operant strategies I (using attention and praise to increase coping), 4) operant strategies II (using rewards to increase positive coping and reach school goals), 5) modeling, 6) lifestyle, 7) communication, 8) relapse prevention.
  Interventions: Behavioral: Web-based CBT (Web-MAP)

INTERVENTIONS:
Behavioral: Web-based CBT (Web-MAP) — see arm description

SUMMARY:
The MOCAS Study aims to describe the mechanisms through which sleep deficiency affects youth responses to an online pain self-management intervention over a 6-month period. The study is a single arm trial with repeated measurements using surveys, daily diaries, and actigraphic monitoring.

DETAILED DESCRIPTION:
The study objective is to characterize how sleep deficiency influences youth's ability to engage with, implement, and benefit from pain self-management intervention. The investigators will recruit a cohort of 80 youth, ages 12 to 17 years, with chronic musculoskeletal, head, or abdominal pain into a single arm trial conducted at one site. Assessments will occur at baseline, immediately after intervention, and repeated at 3 months post-intervention. Mediators will be assessed at mid-treatment (4 weeks). All youth will receive an 8-week internet-delivered pain self-management intervention (WebMAP). Following the recommended Common Data Elements for self-management three self-management processes are measured including patient activation, pain self-efficacy, and self-management skills, and patient-reported outcomes of health (global health, fatigue) and pain (pain symptoms, pain-related disability). Positive and negative affect and executive function are assessed as potential mediators. Sleep deficiency is comprehensively assessed with subjective measures, daily sleep logs, and ambulatory actigraphy monitoring to measure disrupted sleep, amount of sleep, sleep quality, and insomnia symptoms.

ELIGIBILITY:
Inclusion Criteria:

* 12-17 years old
* Has chronic pain (for at least 3 months)
* Has internet access/email address

Exclusion Criteria:

* Diagnosis of a serious, comorbid health condition (e.g. cancer, arthritis, cystic fibrosis, lupus, etc.)
* Parent/adolescent doesn't speak English
* Active psychosis/suicidal ideation
* Currently taking stimulating medications
* Diagnosed sleep disorder (sleep apnea or narcolepsy)
* Severe cognitive impairment/unable to read at 5th grade level or complete surveys independently

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 85 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Law EF, Tham SW, Howard W, Ward TM, Palermo TM. Executive Functioning and Self-Management Processes Mediate the Relationship Between Insomnia and Pain-Related Disability. J Pain. 2024 Jan;25(1):273-283. doi: 10.1016/j.jpain.2023.08.010. Epub 2023 Aug 24. PMID 37633572
- [Derived] de la Vega R, Palermo TM. Mediating Role of Treatment Perceptions in the Relationship Between Individual Characteristics and Engagement With a Digital Psychological Intervention for Pediatric Chronic Pain: Secondary Data Analysis. JMIR Pediatr Parent. 2023 Mar 6;6:e42399. doi: 10.2196/42399. PMID 36877543
- [Derived] Palermo TM, Law EF, Kim A, de la Vega R, Zhou C. Baseline Sleep Disturbances Modify Outcome Trajectories in Adolescents With Chronic Pain Receiving Internet-Delivered Psychological Treatment. J Pain. 2022 Jul;23(7):1245-1255. doi: 10.1016/j.jpain.2022.03.003. Epub 2022 Mar 10. PMID 35283268

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participant gave consent for did not complete the pre-treatment assessment
Period: Baseline
Arm/Group | Web-based CBT (Web-MAP)
Started | 85
Completed | 85
Not Completed | 0
Period: Post-Treatment
Arm/Group | Web-based CBT (Web-MAP)
Started | 85
Completed | 77
Not Completed | 8
Not completed — Declined due to lack of time/interest or could not be reached | 3
Not completed — Withdrawal by Subject | 5
Period: Follow-up
Arm/Group | Web-based CBT (Web-MAP)
Started | 80
Completed | 73
Not Completed | 7
Not completed — Declined due to lack of time/interest or could not be reached | 7

BASELINE CHARACTERISTICS:
Arm/Group | Web-based CBT (Web-MAP)
Number analyzed (Participants) | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 85
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.5 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 72
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 64
  More than one race | 16
  Unknown or Not Reported | 1
Parent education [Count of Participants; unit: Participants]
  High school or less | 4
  College or vocational school | 60
  Graduate or professional school | 20
  Not reported | 1
Annual household income [Count of Participants; unit: Participants]
  $49,999 or less | 24
  $50,000 - $99,999 | 25
  $100,000 or more | 35
  Not reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity Ratings
Description: Pain intensity will be measured using the 11-point Numerical Rating Scale (NRS) completed by children via daily diary assessments over a 7-day period. Scores range from 0 = no pain to 10 = worst pain imaginable. Scores are averaged at each timeframe with higher scores indicating higher pain intensity.
Time Frame: Baseline, 12 weeks (post-treatment), 6 months (follow-up)
Population: At Post-Treatment 3 subjects declined to participate or could not be reached, and 5 subjects withdrew from the study. At Follow-up, of the remaining 80 enrolled participants 7 declined to participate or could not be reached.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Web-based CBT (Web-MAP)
Number analyzed (Participants) | 85
score on a scale
  Baseline | 5.86 (1.66)
  Post-Treatment: number analyzed (Participants) | 77
  Post-Treatment | 5.64 (1.54)
  Follow-up: number analyzed (Participants) | 73
  Follow-up | 5.45 (1.66)

2. Primary Outcome: Pain-related Disability
Description: The Child Activity Limitations Interview (CALI-9) is a daily diary validated to assess perceived difficulty in completing 9 daily activities as a measure of pain-related disability. Responses are rated on a 5-point scale (0-4), summed, and transformed to a 0-100 scale, with higher scores indicating greater perceived difficulty with activities. Youth will provide ratings daily for 7 days on their online diaries at each assessment period. Mean total activity limitations across the reporting period is used in analyses, with higher scores indicating greater disability.
Time Frame: Baseline, 12 weeks (post-treatment), 6 months (follow-up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Web-based CBT (Web-MAP)
Number analyzed (Participants) | 85
score on a scale
  Baseline | 48.33 (21.84)
  Post-Treatment: number analyzed (Participants) | 77
  Post-Treatment | 44.48 (22.52)
  Follow-up: number analyzed (Participants) | 73
  Follow-up | 44.45 (23.40)

3. Secondary Outcome: Fatigue
Description: Children will complete ratings of fatigue on the PedsQL Multidimensional Fatigue Scale, which yields three scores for general fatigue, cognitive fatigue, and sleep-rest fatigue. Scores range from 0-100, where higher scores indicate fewer problems with fatigue. It has been widely used in many pediatric chronic health conditions demonstrating strong reliability and validity.
Time Frame: Baseline, 12 weeks (post-treatment), 6 months (follow-up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Web-based CBT (Web-MAP)
Number analyzed (Participants) | 85
score on a scale
  Baseline | 44.58 (18.24)
  Post-Treatment: number analyzed (Participants) | 77
  Post-Treatment | 48.71 (15.70)
  Follow-up: number analyzed (Participants) | 73
  Follow-up | 47.79 (18.94)

4. Secondary Outcome: Global Health
Description: Global health will be assessed by child self report with the PROMIS pediatric global health scale, a 7-item measure summarizing a child's physical, mental, and social health into a single score. The seven items are rated on a 1-5 scale based on their frequency over the past week. Raw scores are then transformed to a T-Score metric allowing for comparisons to a general (norm) population with mean of 50 and standard deviation of 10. Higher scores mean that the child's global health is more positive.
Time Frame: Baseline, 12 weeks (post-treatment), 6 months (follow-up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Web-based CBT (Web-MAP)
Number analyzed (Participants) | 85
score on a scale
  Baseline | 34.84 (7.38)
  Post-Treatment: number analyzed (Participants) | 77
  Post-Treatment | 36.87 (8.45)
  Follow-up: number analyzed (Participants) | 73
  Follow-up | 38.04 (8.67)

5. Secondary Outcome: Number of Treatment Modules Completed
Description: Measured as the number of pain self-management modules completed by each participant during the intervention period ranging from 0 to 8 modules. Module completion was categorized as no exposure with 0 modules completed vs some exposure with 1-8 modules completed. Module usage information is obtained from the administrative database of the internet program and is stored in real time.
Time Frame: 12 weeks (post-treatment)
Population: Number of treatment modules completed by those completing intervention period
Measure: Count of Participants; unit: Participants
Arm/Group | Web-based CBT (Web-MAP)
Number analyzed (Participants) | 77
Participants
  0 modules completed | 5
  1-8 modules completed | 72

6. Secondary Outcome: Treatment Acceptability
Description: Measured using the Treatment Evaluation Inventory (TEI) completed via teen report, which includes 9 items that are rated on a 5 point likert scale (1-5) where higher scores indicate greater treatment acceptability. Individual scores are summed for a total ranging from 9 to 45, and scores over 37 indicate moderate treatment acceptability.
Time Frame: 12 weeks (post-treatment)
Population: Teen report of treatment acceptability at post-treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Web-based CBT (Web-MAP)
Number analyzed (Participants) | 77
score on a scale | 31.24 (5.60)

ADVERSE EVENTS:
Time Frame: Through study completion and follow-up (average of 6 months)
Description: Standard definitions used in clinicaltrials.gov
Arm/Group | Web-based CBT (Web-MAP)
All-Cause Mortality (participants affected / at risk) | 0/85
Serious Adverse Events (participants affected / at risk) | 0/85
Other Adverse Events (participants affected / at risk) | 0/85

LIMITATIONS AND CAVEATS:
Findings may not generalize to more demographically diverse samples, and patients with specific pain conditions.

Can't determine mediators of treatment effects since it was a single arm trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-02): https://cdn.clinicaltrials.gov/large-docs/62/NCT04043962/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-03): https://cdn.clinicaltrials.gov/large-docs/62/NCT04043962/ICF_001.pdf